CLINICAL TRIAL: NCT03432104
Title: Evaluation of Absorption and Metabolism of Phenolic Compounds From Oxxynea®, a Blend of Fruit and Vegetable Extracts, in Human Healthy Volunteers: a Randomized, Double-blind, Cross-over Trial
Brief Title: Evaluation of Bioavailability of Phenolic Compounds From Oxxynea®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OXCT2018
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Oxxynea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): This arm receives 1 x 450 mg-capsule of Oxxynea®, a blend of polyphenol-rich fruit and vegetable extracts
  Interventions: Dietary Supplement: Oxxynea®; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): This arms receives 1 x 450 mg-capsule of Placebo, containing maltodextrin only
  Interventions: Dietary Supplement: Oxxynea®; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oxxynea® — Oxxynea® is a blend of polyphenol-rich extracts from olive, grape, pomegranate, green tea, grapefruit, orange and blueberry. Dosage is 1 x 450 mg-capsule.
Dietary Supplement: Placebo — Placebo product is 100% maltodextrin. Dosage is 1 x 450 mg-capsule of identical appearance than the verum capsule.

SUMMARY:
The aim of this study is to evaluate bioavailability and pharmacokinetics of phenolic compounds from Oxxynea®, a blend of fruit and vegetable extracts, in healthy volunteers, during a randomized, double-blind and cross-over trial. After a single dose supplementation, both metabolic profile and urinary excretion will be determined over a 48h-period by means of High-Performance Liquid Chromatography coupled with a tandem mass spectrometry (HPLC-MS) to identify and quantify phenolic metabolites. In parallel, post-prandial potential anti-oxidative and anti-glycemic properties of Oxxynea® will be determined in blood, following consumption of a cafeteria-type breakfast.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Agreement to adhere to diet considerations

Exclusion Criteria:

* Smoking
* Pregnancy / Lactation
* Current use of any medication or food supplement
* Known allergic reaction to components of the supplement/placebo

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of phenolic metabolites after acute ingestion of the supplement/placebo | 0h, 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 24h post-ingestion
  Plasma samples will be collected in EDTA tubes in baseline before supplement/placebo intake (0h) and up to 24h according to the time frame. Plasma metabolites will be identified and quantified by HPLC-MS.

SECONDARY OUTCOMES:
Change in urine phenolic metabolites excretion after acute ingestion of the supplement/placebo | Baseline (12h pre-ingestion), 0-3h, 3-6h, 6-10h, 10-14h, 14-24h, 24-32h, 32-48h post-ingestion
  Urine samples will be collected in baseline (12h pre-ingestion) and up to 48h according to the time frame. Urine metabolites will be identified and quantified by HPLC-MS.
Change in total circulating antioxidant defences after acute ingestion of the supplement/placebo | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 24h post-ingestion
  Red blood cell (RBCs) samples will be collected in EDTA tubes in baseline before supplement/placebo intake (0h), 1h post-ingestion and following a cafeteria-type breakfast, and up to 24h according to the time frame.
  RBCs will be submitted to the KRL (Kit Radicaux Libres) test which consists in inducing a free-radical attack to RBCs and to follow hemolysis. Results will be expressed as the time required to reach 50% of maximal hemolysis.
Change in post-prandial glycemia | 0h, 1h, 2h, 3h, 4h, 5h, 6h post-ingestion
  Glycemia will be measured in a fasted state in baseline before supplement/placebo intake (0h), 1h post-ingestion and following a cafeteria-type breakfast, and up to 6h according to the time frame.
Change in post-prandial insulinemia | 0h, 1h, 2h, 3h, 4h, 5h, 6h post-ingestion
  Insulinemia will be measured in a fasted state in baseline before supplement/placebo intake (0h), 1h post-ingestion and following a cafeteria-type breakfast, and up to 6h according to the time frame.
Change in sleepiness during the day | 0h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 10h post-ingestion
  Change in sleepiness will be assessed using the Stanford Sleepiness Scale (SSS), a 7-point self-rating scale. The scale is used to track overall alertness during the day. At each point of the time frame, volunteers will be asked to rate their feelings of sleepiness from 1 to 7 according to the following descriptors:
  1. Feeling active, vital, alert, or wide awake
  2. Functioning at high levels, but not at peak; able to concentrate
  3. Awake, but relaxed; responsive but not fully alert
  4. Somewhat foggy, let down
  5. Foggy; losing interest in remaining awake; slowed down
  6. Sleepy, woozy, fighting sleep; prefer to lie down
  7. No longer fighting sleep, sleep onset soon; having dream-like thoughts

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Alcaraz Ramon, Principal Investigator — UCAM (Universidad Catolica San Antonio de Murcia)
Locations (1):
- UCAM (Universidad Catolica San Antonio de Murcia), Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided